CLINICAL TRIAL: NCT06982820
Title: A Prospective, Randomized, Double-blind, Controlled Study to Produce Guidelines for Integrating Prism for MDD Therapy (Reward System [RS] Upregulation) and to Demonstrate Its Superiority Over Sham Therapy
Brief Title: Self Neuro-modulation Therapy for Major Depressive Disorder (MDD) With Anhedonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GrayMatters Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLP015
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder (MDD); Anhedonia; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia; Depression

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blind, controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind: neither participants nor clinicians assessing them will have information regarding the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active arm (Active Comparator): Participants randomized into the Active arm will receive reward system EEG-fMRI pattern (RS-EFP) Neuro Feedback (NF) Prism training as an adjunct to SOC.
  Interventions: Device: Prism Training
- Sham arm (Sham Comparator): Participants randomized into the Sham arm will receive a Sham EFP-NF training with the same schedule as the active arm, adjunct to SOC.
  Interventions: Device: Prism Training

INTERVENTIONS:
Device: Prism Training — Participants will complete 20 Prism training sessions. The Prism training sessions take place twice a week over a 10-week period, with a minimum of one night of sleep between sessions. Participants will also receive two single booster sessions, 4 weeks and 8 weeks after their last NF session completed.
  Other Names: Sham Training

SUMMARY:
The purpose of this research is to learn more about a new treatment for individuals with Major Depressive Disorder (MDD) with heightened symptoms of anhedonia (i.e. loss of pleasure or interest in activities). The treatment is called Prism, and it is a software device intended for a novel form of neurofeedback training to be used in a clinic setting.

During this study, the subject will use different techniques to measure brain activities, including magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
The study is comprised of the Screening Visit, Baseline Assessment, Pre-training Visit, 20 NF Training Visits (two training visits per week over 10 weeks), two Booster NF Training Visits (Week 16, and Week 20, and the 3-Month Follow-up Assessment Visit (Week 24).

Participants will receive 20 NF sessions.

The study will test the following hypothesis:

* H0: M(Anhedonic)RS-EFP = M(Anhedonic)Sham-EFP
* H1: M(Anhedonic)RS-EFP ≠ M(Anhedonic)Sham-EFP

Where:

M(Anhedonic)RS-EFP and M(Anhedonic)Sham-EFP are the mean changes from baseline HDRS-17 score in the Active and Sham arms of the Anhedonic MDD participants.

*HDRS-21 is administered for cluster analysis

ELIGIBILITY:
Inclusion Criteria:

1. Primary Diagnosis of MDD with Anhedonia, established according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM5TR) - HDRS-17 score of ≥20, SHAPS-C score of ≥25.
2. Fluency in written and spoken English.
3. Able intellectually to understand the instructions
4. Ability to give signed, informed consent either written or electronic (via REDCap eConsent).
5. Normal or corrected-to-normal vision and hearing.
6. Ability to adhere to the study schedule.
7. Completed at least one antidepressant treatment course at an adequate dose and duration in the current episode per the ATRQ.

Exclusion Criteria:

1. Contraindications to MRI (e.g., metal in the body, claustrophobia).
2. Any suicidal behavior in the past 1 year (i.e., actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior) assessed using Columbia -Suicide Severity Rating Scale (C-SSRS) prior to screening and during the screening period.
3. Diagnosis for current moderate or severe substance or alcohol use disorder (SUD/AUD) within the past month (as defined in DSM-5-substance use disorder).
4. Any unstable medical condition, as per the clinical judgement of the investigator.
5. Any change in, or initiation of, fluoxetine within the past 8 weeks or of other SSRIs/SNRIs antidepressants, bupropion, stimulants, or other psychiatric medications within the past 4 weeks.
6. Recent initiation (within the past 2 months) of psychotherapy; continuation of established maintenance supportive therapy will be permitted.
7. Enrollment in another therapeutic clinical study at screening or within 2 months prior to screening or intended enrollment within the duration of this study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
HDRS-21 | Change from baseline to week 12 (post training visit)
  Hamilton Rating Scale for Depression - the maximum score is 64. A score above 20 is considered a severe depression.

SECONDARY OUTCOMES:
SHAPS-C | Change from baseline to week 12 (post-training visit)
  Snaith-Hamilton-Pleasure scale - is a 14- item self-administered measure of anhedonia symptoms.
HDRS-21 | Change from baseline to 3-month FU visit
  Hamilton Rating Scale for Depression - the maximum score is 64. A score above 20 is considered a severe depression.
CGI-I | Change from baseline to week 12 (post-training visit)
  Clinical global impression - The 7-point CGI-I scale rates improve with a (1) representing a very much improved' patient and (7) representing a patient who has become 'very much worse' due to treatment. The rating (4) represents a patient displaying no change from the treatment.
CGI-I | Change from week 12 to 3-Month follow-up Assessment
  Clinical global impression - The 7-point CGI-I scale rates improve with a (1) representing a very much improved' patient and (7) representing a patient who has become 'very much worse' due to treatment. The rating (4) represents a patient displaying no change from the treatment.
PHQ-9 | Change from baseline to week 12 (post-Training visit)
  Patient Health Questionnaire-9 - The PHQ-9 is a nine-item depressive symptom diagnostic tool.

CONTACTS AND LOCATIONS:
Overall Officials: Aron Tendler, MD, Study Director — GrayMatters Health
Locations (2):
- United States (2):
  - Novus Psychiatry, Tuscaloosa, Alabama
  - Butler Hospital, Providence, Rhode Island